CLINICAL TRIAL: NCT00500149
Title: A Phase IIIb, Randomized, Double-Blind, Multi-Center, Placebo- Controlled, Dose-Optimization, Cross-Over, Analog Classroom Study to Assess the Time of Onset of Vyvanse (Lisdexamfetamine Dimesylate) in Pediatric Subjects Aged 6-12 With Attention-Deficit/Hyperactivity Disorder
Brief Title: A Classroom Study to Assess the Time of Onset of Vyvanse (Lisdexamfetamine Dimesylate) in Pediatric Subjects Aged 6-12 With Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-311
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2009-06-05 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Vyvanse (lisdexamfetamine dimesylate)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vyvanse (lisdexamfetamine dimesylate) — Following completion of the open-label dose optimization period and successful titration to an optimal dose of Vyvanse™, subjects will take their optimized dose of Vyvanse™ (30, 50 or 70 mg/day).
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The primary objective of this study is to assess the time of onset of Vyvanse compared to placebo, in the analog classroom as measured by the Swanson, Kotkin, Agler, M. Flynn and Pelham (SKAMP) deportment scale in children (aged 6-12) diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female aged 6-12 years inclusive at the time of consent.
2. Females of Child-bearing Potential (FOCP) must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to comply with any applicable contraceptive requirements of the protocol.
3. Primary diagnosis of ADHD: combined sub-type or predominantly hyperactive impulsive sub-type based on a detailed psychiatric evaluation.
4. Subject has a baseline ADHD-RS-IV score ≥ 28.
5. Intelligent Quotient (IQ) score of 80 or above on the Kaufman Brief Intelligence Test (KBIT).
6. Subject must be able to complete at least the Basic Test of the PERMP assessment.

Exclusion Criteria:

1. Subject has a current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as Post Traumatic Stress Disorder (PTSD), psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder
2. Subject has Conduct Disorder.
3. Subject has a documented allergy, hypersensitivity or intolerance to amphetamines.
4. Subject has failed to respond to one or more adequate courses (dose and duration) of amphetamine therapy.
5. The subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-IV-TR criteria.
6. Subject weighs less than 50 pounds (22.7kg).
7. Subject is significantly overweight
8. Subject had a history of seizures during the last two years (exclusive of febrile seizures), a tic disorder, a current diagnosis and/or family history of Tourette's Disorder.
9. Subject has any reported history of abnormal thyroid function.
10. Subject has taken another investigational drug or taken part in a clinical trial within the last 30 days prior to Screening.
11. Subject has a known history of structural cardiac abnormality, as well as any other condition(s) that may affect cardiac performance.
12. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments
13. Subject is taking other medications that have central nervous system (CNS) effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics (bronchodilators are not exclusionary).
14. The female subject is pregnant or lactating.
15. Subject is well controlled on their current ADHD medication with acceptable tolerability.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2007-06-13 (Actual); Primary Completion 2007-12-05 (Actual); Study Completion 2007-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (9):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Univ. of CA, Irvine Child Development Center, Irvine, California
  - Shire Clinical Research Site, Wildomar, California
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Center for Psychiatry & Behavioral Medicine Inc, Las Vegas, Nevada
  - Duke Child & Family Study Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Shire Clinical Research Site, Houston, Texas
  - Shire Clinical Research Site, Lubbock, Texas

REFERENCES:
- [Result] Wigal SB, Kollins SH, Childress AC, Squires L; 311 Study Group. A 13-hour laboratory school study of lisdexamfetamine dimesylate in school-aged children with attention-deficit/hyperactivity disorder. Child Adolesc Psychiatry Ment Health. 2009 Jun 9;3(1):17. doi: 10.1186/1753-2000-3-17. PMID 19508731
- [Result] Wigal SB, Kollins SH, Childress AC, Adeyi B. Efficacy and tolerability of lisdexamfetamine dimesylate in children with attention-deficit/hyperactivity disorder: sex and age effects and effect size across the day. Child Adolesc Psychiatry Ment Health. 2010 Dec 14;4:32. doi: 10.1186/1753-2000-4-32. PMID 21156071
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 129 subjects were enrolled for dose optimization phase, 12 discontinued, and 117 were randomized to the cross-over phase.
Pre-assignment Details: The study consisted of an open-label dose-optimization phase (4 weeks), followed by a randomized, placebo-controlled, 2-way crossover phase (1 week each).
Groups:
- Vyvanse First: Vyvanse was dosed orally once daily at either 30, 50 or 70 mg (depending on the outcome of the dose optimization phase)for 1 week in the first intervention and matching placebo was given orally once daily for 1 week in the second intervention
- Placebo First: Matching placebo was given orally once daily for 1 week in the first intervention and Vyvanse was dosed orally once daily at either 30, 50 or 70 mg (depending on the outcome of the dose optimization phase)for 1 week in the second intervention
Period: Enrolled (Dose-optimization Phase)
Arm/Group | Vyvanse First | Placebo First
Started | 129 | 0
Completed | 117 | 0
Not Completed | 12 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 8 | 0
Not completed — Protocol Violation | 1 | 0
Period: First Intervention (Cross-over Phase)
Arm/Group | Vyvanse First | Placebo First
Started | 58 | 59
Completed | 56 | 57
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention (Cross-over Phase)
Arm/Group | Vyvanse First | Placebo First
Started | 56 | 57
Completed | 54 | 57
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 129
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 98
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 129

OUTCOME MEASURES:

1. Primary Outcome: Onset of Effect of Vyvanse
Description: The onset of effect will be defined as the first assessment time showing statistical significance between Vyvanse and placebo as measured by the Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Deportment scale. The degree of impairment is rated from 0 (normal) to 6 (maximal).
Time Frame: Evaluations were conducted at 1.5, 2.5, 5.0, 7.5, 10.0, 12.0, and 13.0 hours post-dose.
Population: Analysis on the intention-to-treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Vyvanse: Lisdexamfetamine dimesylate (LDX)
- Placebo: Matching placebo
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 113 | 113
scores on a scale
  1.5 hours | 0.70 (0.09) | 1.14 (0.09)
  2.5 hours | 0.45 (0.09) | 1.42 (0.09)
  5 hours | 0.44 (0.10) | 1.60 (0.10)
  7.5 hours | 0.54 (0.09) | 1.56 (0.09)
  10 hours | 0.60 (0.09) | 1.43 (0.09)
  12 hours | 0.90 (0.10) | 1.41 (0.10)
  13 hours | 1.05 (0.10) | 1.31 (0.10)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 1.5 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — The primary efficacy variable will be onset of effect, which will be determined from the results of inferential analyses across multiple time points. No adjustment will be made to the levels of significance as a result of the multiple comparisons; Using a linear mixed model that includes sequence, period, and treatment group as fixed effects and subject-within-sequence as a random effect
Statistical Analysis 2: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 2.5 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 5.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 7.5 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 10.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 12.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 13.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Duration of Effect of Vyvanse
Description: Duration of effect will be defined as the first time point at which there is a non-significant difference between Vyvanse and placebo after a time point at which there is a significant difference between the two treatment groups as measured by SKAMP Deportment Scores. The degree of impairment is rated from 0 (normal) to 6 (maximal).
Time Frame: Evaluations were conducted at 1.5, 2.5, 5.0, 7.5, 10.0, 12.0, and 13.0 hours post-dose.
Population: Analysis on intention-to-treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 113 | 113
scores on a scale
  1.5 hours | 0.70 (0.09) | 1.14 (0.09)
  2.5 hours | 0.45 (0.09) | 1.42 (0.09)
  5 hours | 0.44 (0.10) | 1.60 (0.10)
  7.5 hours | 0.54 (0.09) | 1.56 (0.09)
  10 hours | 0.60 (0.09) | 1.43 (0.09)
  12 hours | 0.90 (0.10) | 1.41 (0.10)
  13 hours | 1.05 (0.10) | 1.31 (0.10)
Statistical Analysis 1: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 1.5 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 2.5 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 5.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 7.5 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 10.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 12.0 hours post-dose; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Vyvanse vs Placebo; Statistical analysis of SKAMP scores at 13.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: The Randomized Population is defined as all subjects who are randomized and received at least one dose of study medication during the Cross-Over Phase of the study.
Arm/Group | Vyvanse | Placebo
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/115
Other Adverse Events (participants affected / at risk) | 13/115 | 3/115
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vyvanse (N=115) | Placebo (N=115)
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 1
Headache (Nervous system disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after SPONSOR confirms there shall be no multicenter Study publication, the INSTITUTION and/or such PRINCIPAL INVESTIGATOR may publish the results from the INSTITUTION site individually.